CLINICAL TRIAL: NCT07365085
Title: Whole Versus Segmented In-House 3D Mandibular Guides for Mandibular Reconstruction Using Free Fibular Flaps: A Randomized Clinical Trial
Brief Title: Whole vs Segmented 3D Models for Mandibular Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kristaninta Bangun, Kristaninta Bangun, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3DFFF
Record Dates: First submitted 2026-01-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: 3d Printing; Facial Symmetry; Free Fibular Flap; 3d Model; Mandibular Reconstruction
Keywords: 3d printing; facial symmetry; free fibular flap; 3d model; mandibular reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEGMENTED MODEL (Experimental): Segmented 3D Mandibular Model.
  Interventions: Device: 3D-printed surgical guide - segmented model
- WHOLE MANDIBLE MODEL (Active Comparator): Whole 3D Mandibular Model.
  Interventions: Device: 3D-printed surgical guide - whole mandible model

INTERVENTIONS:
Device: 3D-printed surgical guide - segmented model — In this technique, a 3D scan of the patient's mandible was isolated, the defect excised, mimicking post-surgical resection mandible. Then, the 3D scan of the patient's fibula was isolated and arranged into segments to match the post-resection defect of the mandible. The final result would resemble the patient's mandible after reconstruction with free fibular flap.
  Arms: SEGMENTED MODEL
Device: 3D-printed surgical guide - whole mandible model — In this technique, the patient's mandibular anatomy was segmented from the preoperative 3D scan, and the diseased portion of the mandible was digitally removed. The unaffected hemimandible was then mirrored across the sagittal plane to generate a symmetrical, anatomically normal mandibular contour. When the defect extended beyond the midline, a standardized normal mandibular model was digitally trimmed and adapted to the patient's anatomy by adjusting the intercondylar distance and mandibular curvature. The finalized model was positioned within the patient's mandibular fossa to ensure accurate anatomical alignment and optimal fit.
  Arms: WHOLE MANDIBLE MODEL

SUMMARY:
Three-dimensional (3D) printing is increasingly used in surgery to help doctors plan and perform complex operations with greater accuracy. In this study, the investigators used 3D-printed jaw models to assist in rebuilding the lower jaw (mandible) after tumor removal, using bone taken from the lower leg in a procedure called a free fibular flap.

The investigators compared two types of 3D-printed mandibular guides. One used a complete model of the patient's healthy mandible to guide reconstruction, while the other rebuilt the jaw by dividing the leg bone into planned segments and fitting them precisely into the jaw defect. All 3D design and printing were performed in-house by the surgical team using free computer software.

After surgery, the investigators evaluated facial symmetry using standardized photographs taken before surgery and three months afterward. Both techniques helped surgeons achieve good reconstruction results. However, the segmented model produced more consistent facial symmetry, while results from the whole-mandible model varied more between patients.

Overall, this study shows that in-house 3D printing is a practical and affordable tool for jaw reconstruction surgery. Although both approaches were effective, segmented models may offer more reliable results. Larger studies are needed to confirm these findings and improve future patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing segmental mandibular reconstruction with a free fibular flap.
2. Mandibular defects resulting from benign tumors, malignant tumors, trauma, or osteonecrosis requiring reconstruction.
3. Availability of preoperative high-resolution CT imaging suitable for virtual surgical planning and 3D modeling.
4. Agreed and signed the consent forms

Exclusion Criteria:

1. Contraindications to free fibular flap harvest (e.g., significant peripheral vascular disease, prior fibular surgery).
2. History of previous mandibular reconstruction or major maxillofacial surgery altering baseline anatomy.
3. Preexisting severe facial asymmetry unrelated to the mandibular defect.
4. Inadequate imaging data or incomplete medical records.
5. Incomplete or poor-quality postoperative photographs preventing accurate asymmetry measurement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
FACIAL SYMMETRY | From enrollment to 1 month postoperatively
  Postoperative assessment of facial symmetry was performed using clinical photographs and plain radiograph of the head (AP) taken 1 month after surgery. The facial asymmetry index (AI) was calculated using the formula:
  AI (%) = (R - L)/(R + L) × 100%, based on cephalometric landmarks including sella-nasion (Sn), angle of the mouth (Am), and soft tissue pogonion (Po) (Figure 3), in accordance with the method described by Nakamura et al.⁴. This index represents the proportional difference between the right and left sides of each landmark relative to total facial width, expressed as a percentage. Higher AI values indicate greater facial asymmetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Central Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Probst FA, Liokatis P, Mast G, Ehrenfeld M. Virtual planning for mandible resection and reconstruction. Innov Surg Sci. 2023 Dec 6;8(3):137-148. doi: 10.1515/iss-2021-0045. eCollection 2023 Sep. PMID 38077486
- [Result] Barr ML, Haveles CS, Rezzadeh KS, Nolan IT, Castro R, Lee JC, Steinbacher D, Pfaff MJ. Virtual Surgical Planning for Mandibular Reconstruction With the Fibula Free Flap: A Systematic Review and Meta-analysis. Ann Plast Surg. 2020 Jan;84(1):117-122. doi: 10.1097/SAP.0000000000002006. PMID 31633539
- [Result] Davies JC, Chan HHL, Jozaghi Y, Goldstein DP, Irish JC. Analysis of simulated mandibular reconstruction using a segmental mirroring technique. J Craniomaxillofac Surg. 2019 Mar;47(3):468-472. doi: 10.1016/j.jcms.2018.12.016. Epub 2018 Dec 30. PMID 30661926
- [Result] Nakamura T, Okamoto K, Maruyama T. Facial asymmetry in patients with cervicobrachial pain and headache. J Oral Rehabil. 2001 Nov;28(11):1009-14. doi: 10.1046/j.1365-2842.2001.00766.x. PMID 11722716
- [Result] Kargilis DC, Xu W, Reddy S, Ramesh SSK, Wang S, Le AD, Rajapakse CS. Deep learning segmentation of mandible with lower dentition from cone beam CT. Oral Radiol. 2025 Jan;41(1):1-9. doi: 10.1007/s11282-024-00770-6. Epub 2024 Aug 14. PMID 39141154
- [Result] Bosc R, Hersant B, Carloni R, Niddam J, Bouhassira J, De Kermadec H, Bequignon E, Wojcik T, Julieron M, Meningaud JP. Mandibular reconstruction after cancer: an in-house approach to manufacturing cutting guides. Int J Oral Maxillofac Surg. 2017 Jan;46(1):24-31. doi: 10.1016/j.ijom.2016.10.004. Epub 2016 Nov 2. PMID 27815013
- [Result] Chiu YT, Liao YF. Is cleft severity related to maxillary growth in patients with unilateral cleft lip and palate? Cleft Palate Craniofac J. 2012 Sep;49(5):535-40. doi: 10.1597/10-044. Epub 2010 Dec 23. PMID 21214323